CLINICAL TRIAL: NCT00227097
Title: Implication of Patient in the Making Ready of Recommendations for the Antivitamin K's Gestion in Case of Thrombosis Embolic Venous's Illness. Randomised Study for Clinical Validation.
Brief Title: Educ'Avk: Recommendations for the Antivitamin K's Gestion
Status: Terminated | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Other Study IDs: DCIC 02 03
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2006-07-07 (Estimated); Status verified 2006-07

CONDITIONS: AVK Treatment
Keywords: therapeutic education; thrombi embolic disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Education Notebook for anticoagulant treatment

SUMMARY:
The objective of the project "Educ'Avk", is to document the efficacy of a strategy combining a specific follow up-notebook and education of attending patient with a pedagogic support, comparatively to an usual education on the impact of clinical events at three months (minor or major hemorrhagic events + recurrence of thrombi-embolic's disease).

DETAILED DESCRIPTION:
Standard strategies for the implementation of recommendations are exclusively focused on practitioners. But often they do not appear to be effective (insufficient time accorded per patient, lack of training…).

However some qualitative surveys have shown the benefit of a greater role on the part patient in the process of transmitting recommendations through the practitioner.

In this study, patient education is begun by the angiologist or a pharmacy student under the responsibility of the hospital investigator. Follow-up is realized by the patient's general practitioner.

More patient involvement in the realization of the recommendations could increase the proportion of practitioners who follow the recommendations and decrease the iatrogenicity of antivitamin K (AVK).

ELIGIBILITY:
Inclusion Criteria:

* Able to receive benefit sanitary educational act
* Able to be followed up during three months
* Acute episode of a venous's thrombi embolic illness (venous's thrombosis distal or proximal deep and/or lung embolism)
* A.V.K. treatment for a period of at least three months
* Return to residence (included return to retreat residence no medicalize)
* Informed consent form signed

Exclusion Criteria:

* Distal venous thrombosis limited muscular vein without lung embolism
* Contra-indication of to an A.V.K. treatment
* Difficult comprehension of the french language
* Trouble of visual acuity
* Trouble of superior function incompatible with an educational's act sanitary
* Psycho-social instability incompatible with a regular follow-up of three months (without fixed residence, addictive lapsed)
* Impossibility to return to residence (the return in retreat residence no medicalize is considered as a return to residence)
* Psychiatric pathology not compensated
* Life expectancy less than three months
* Refusal of participation in the study
* Participation in another clinical study
* Anterior inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-12; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc BOSSON, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Cardiovascular Departement - University Hospital of Grenoble - BP 217, La Tronche, Grenoble Cédex 9, France

REFERENCES:
- [Background] Gratacap-Cavallier B, Bosson JL, Morand P, Dutertre N, Chanzy B, Jouk PS, Vandekerckhove C, Cart-Lamy P, Seigneurin JM. Cytomegalovirus seroprevalence in French pregnant women: parity and place of birth as major predictive factors. Eur J Epidemiol. 1998 Feb;14(2):147-52. doi: 10.1023/a:1007450729633. PMID 9556173
- [Background] Bertrand D, Francois P, Bosson JL, Fauconnier J, Weil G. Quality assessment of discharge letters in a French university hospital. Int J Health Care Qual Assur Inc Leadersh Health Serv. 1998;11(2-3):90-5. doi: 10.1108/09526869810213019. PMID 10185321
- [Background] Mezin P, Payen JF, Bosson JL, Brambilla E, Stieglitz P. Histological support for the difference between malignant hyperthermia susceptible (MHS), equivocal (MHE) and negative (MHN) muscle biopsies. Br J Anaesth. 1997 Sep;79(3):327-31. doi: 10.1093/bja/79.3.327. PMID 9389850
- [Background] Payen JF, Bosson JL, Bourdon L, Jacquot C, Le Bas JF, Stieglitz P, Benabid AL. Improved noninvasive diagnostic testing for malignant hyperthermia susceptibility from a combination of metabolites determined in vivo with 31P-magnetic resonance spectroscopy. Anesthesiology. 1993 May;78(5):848-55. doi: 10.1097/00000542-199305000-00007. PMID 8489056
- [Background] Vermont J, Bosson JL, Francois P, Robert C, Rueff A, Demongeot J. Strategies for graphical threshold determination. Comput Methods Programs Biomed. 1991 Jun;35(2):141-50. doi: 10.1016/0169-2607(91)90072-2. PMID 1914452